CLINICAL TRIAL: NCT02730780
Title: The Natriuretic Peptide System in African-Americans.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Deepak Gupta, Principal Investigator, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 151943
Record Dates: First submitted 2016-03-29; First posted 2016-04-06 (Estimated); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Healthy; Prehypertension
MeSH Terms: conditions — Prehypertension | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- African-American (Other): 40 healthy African-American subjects will be enrolled and each will undergo study procedures at 4 separate visits, with each visit occurring 7-days apart. After a baseline visit, the subject will begin either a low-salt or high-salt diet, based upon randomization assignment to one of the two following dietary protocols: A) low-salt diet, washout, then high-salt diet; or B) high-salt diet, washout, then low-salt diet. Each dietary or washout period lasts for 7 days.
  Interventions: Dietary Supplement: Low-Salt Diet; Dietary Supplement: High-Salt Diet
- Whites (Other): 40 healthy white subjects will be enrolled and each will undergo study procedures at 4 separate visits, with each visit occurring 7-days apart. After a baseline visit, the subject will begin either a low-salt or high-salt diet, based upon randomization assignment to one of the two following dietary protocols: A) low-salt diet, washout, then high-salt diet; or B) high-salt diet, washout, then low-salt diet. Each dietary or washout period lasts for 7 days.
  Interventions: Dietary Supplement: Low-Salt Diet; Dietary Supplement: High-Salt Diet

INTERVENTIONS:
Dietary Supplement: Low-Salt Diet — The low-salt diet (7 days) will consist of meals, snacks, and sodium free water provided by the study staff.
Dietary Supplement: High-Salt Diet — The high-salt diet (7 days) consists of each subject's usual diet, supplemented each day with 2 bouillon broth packets, which will be provided to the subject by the study staff.

SUMMARY:
This study aims to assess the natriuretic peptide response to dietary salt loading in African-American individuals compared with white individuals.

DETAILED DESCRIPTION:
High blood pressure, or hypertension, is a major cause of heart disease, heart failure, and stroke. Natriuretic peptides are cardiac derived hormones that may protect against hypertension. The classical actions of the natriuretic peptides include natriuresis, vasodilation, and inhibition of the renin-angiotensin-aldosterone system (RAAS), which support a key role for these hormones in blood pressure regulation.

Race based differences exist in the risk and severity of hypertension and cardiovascular disease, with African-American individuals typically being at greater risk compared with white individuals. Nearly half of African-American adults have hypertension, compared with one-third of whites. Additionally, salt-sensitivity denotes the impaired ability to handle a salt load with resulting increases in blood pressure. It is estimated that 75% of hypertensive African-Americans exhibit salt-sensitivity, compared with 35% of hypertensive whites. Why this predilection towards salt-sensitivity exists, particularly among African-American individuals, is not well understood. Thus, establishing the origins of salt retention in African Americans has biologic, preventative, and therapeutic importance, and may provide insight regarding racial differences in cardiovascular risk.

The natriuretic peptide system is the principal counter-regulatory mechanism to salt retention. However, little is known regarding racial differences in the natriuretic peptide system. Recently, it was discovered that African-Americans have lower natriuretic peptide levels compared with whites, raising the possibility that African-Americans individuals can have a relative "natriuretic peptide deficiency" with reduced natriuretic peptide responses to salt loading. However, the prior studies were based on epidemiologic data with individuals on random salt backgrounds. This highlights the need for more detailed physiologic studies, under controlled salt conditions and with standardized assessment of the natriuretic peptide and RAAS and tissue sodium stores.

The aim of this study is to assess the natriuretic peptide response to dietary salt loading in African-American individuals compared with white individuals. This study will test the primary hypothesis that compared with whites, African-American individuals have blunted natriuretic peptide responses to dietary salt loading.

Secondary hypotheses include:

1. Compared with white individuals, African-American individuals have higher baseline tissue sodium content, and
2. Compared with white individuals, African-American individuals have impaired "target organ" responses to salt loading, as manifested by higher blood pressure and increased frequency of salt-sensitive hypertension, decreased urinary sodium excretion, less suppression of plasma renin and serum aldosterone, and lack of increase in left ventricular early diastolic relaxation velocities.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 55 years
* BMI between 18 and <25 kg/m2
* normotensive or pre-hypertensive
* willing to adhere to study diets

Exclusion Criteria:

* prevalent cardiovascular disease or use of medications for cardiovascular disease
* Current or prior history of hypertension or use of blood pressure lowering medications
* Current or prior history of diabetes mellitus or use of anti-diabetic medications
* Prevalent renal disease (eGFR < 60 ml/min/1.73m2), abnormal serum sodium or potassium
* Current or prior smoker
* Current pregnancy
* Current steroid use
* Contraindications to MRI

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
The difference in circulating NT-proANP levels in response to low and high dietary salt. | 4 years

SECONDARY OUTCOMES:
Tissue sodium content | 4 years
  Measured by sodium MRI
Blood pressure | 4 years
Salt-sensitive hypertension | 4 years
  Measured by change in mean arterial pressure
Urinary sodium excretion | 4 years
  Measured from 24 hour urine collection
Myocardial early relaxation velocities | 4 years
  Measured from Echocardiography as tissue Doppler e'
Plasma renin | 4 years
  Physiological parameter
Serum aldosterone | 4 years
  Physiological parameter

CONTACTS AND LOCATIONS:
Overall Officials: Deepak K Gupta, MD, Principal Investigator — Vanderbilt Cardiovascular Medicine
Locations (1):
- Vanderbilt Univeristy, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Gupta DK, de Lemos JA, Ayers CR, Berry JD, Wang TJ. Racial Differences in Natriuretic Peptide Levels: The Dallas Heart Study. JACC Heart Fail. 2015 Jul;3(7):513-519. doi: 10.1016/j.jchf.2015.02.008. Epub 2015 Jun 10. PMID 26071618
- [Background] Gupta DK, Claggett B, Wells Q, Cheng S, Li M, Maruthur N, Selvin E, Coresh J, Konety S, Butler KR, Mosley T, Boerwinkle E, Hoogeveen R, Ballantyne CM, Solomon SD. Racial differences in circulating natriuretic peptide levels: the atherosclerosis risk in communities study. J Am Heart Assoc. 2015 May 21;4(5):e001831. doi: 10.1161/JAHA.115.001831. PMID 25999400